CLINICAL TRIAL: NCT06664840
Title: MyRareDiet™: A Diet Tracking, Monitoring and Optimization mHealth Tool for Patients With Inborn Errors of Metabolism
Brief Title: MyRareDiet A Novel Diet Tracking Tool
Acronym: MRD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: BrightOutcome (Industry); National Urea Cycle Disorder Foundation (Unknown); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Melanie B Gillingham, Professor, Oregon Health and Science University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 1R44HD107766 (NIH); 1R44HD107766 (NIH)
Record Dates: First submitted 2024-10-26; First posted 2024-10-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Urea Cycle Disorder; Propionic Aciduria; Maple Syrup Urine Disease; Methylmalonic Acidemia
MeSH Terms: conditions — Urea Cycle Disorders, Inborn; Propionic Acidemia; Maple Syrup Urine Disease; Methylmalonic acidemia

STUDY DESIGN:
Intervention Model Description: This study is to conduct a validity study to test the agreement between MyRareDiet and the validated interview-based 24-hour diet recall method used in the National Health and Nutrition Examination Survey (NHANES).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MyRareDiet (Experimental): MyRareDiet (MRD) entries: Participants will enter their dietary intake into the MyRareDiet app on a series of three random nonconsecutive days. Participants will receive reminders from both OHSU bionutritionist (via email, phone, or text) and from the MRD system to record their dietary intake on the MRD app for particular randomized days.
  Interventions: Other: MDR diet assessment
- 24 hour recall (Active Comparator): 24-hour diet recalls: A series of three randomized nonconsecutive days of 24-hour food recall interviews by telephone will be completed by trained OHSU Bionutrition personnel to determine nutrient intake. Dietary intake will be evaluated with on Nutrition Data System for Research (NDSR) and Metabolic Pro nutrient databases.
  Interventions: Other: 24 hour recall

INTERVENTIONS:
Other: MDR diet assessment — Participants will record their dietary intake on the MyRareDiet (MRD) app and nutrient content will be assessed to validate MRD compared to a traditional interviewer assessed 24 hour recall.
  Arms: MyRareDiet
Other: 24 hour recall — A trained nutritionist will conduct a telephone multi-pass 24 hour diet recall on 3 randomized nonconsecutive days. The dietary intake will be analyzed using NDSR and metabolic pro and nutrient intake will be compared to the nutrient intake assessed with the MRD app.
  Arms: 24 hour recall

SUMMARY:
The investigators propose to develop and validate MyRareDiet® (MRD) to address an unmet need in the inborn errors of metabolism (IEM) population to assist with dietary management designed to increase adherence and compliance to treatment guidelines, while facilitating the collection of dietary data from individuals with IEM for research purposes.

DETAILED DESCRIPTION:
Inborn errors of metabolism (IEM) are a group of rare genetic disorders that cause a block in a metabolic pathway leading to clinically significant consequences. Most of the disorders are caused by single gene defects that result in a deficiency of a particular enzyme that metabolizes dietary nutrients, eventually causing an accumulation of abnormal metabolites, lack of endogenous production of substances, and/or production of toxic substances that have catastrophic effects on the brain and organs. IEM can lead to developmental and intellectual disabilities, seizures, and, if untreated, coma and death. The majority of the disorders are managed by manipulation and modification of diet alone to reduce toxic metabolites, or with a combination of dietary modification and medications. The complex dietary therapies used in IEM challenge routine dietary recommendations and render diet apps designed for the general public of little utility in these conditions. Additionally, no diet app is developed specifically for the IEM community and meets the rigor required for research, particularly the need to measure specific and multiple amino acids, fats and carbohydrates in the diet to facilitate more study on impact on brain and organs. In IEM, paper diet diaries are often utilized to track food intake and inform patients and their dietitians whether their diets are consistent with the therapy recommendations. These diaries are frequently inadequate in capturing what is actually being consumed due to recall errors and other factors. Novel methods of assessing dietary intake are required to reduce the diet tracking burden, improve accuracy in dietary surveys, and improve diet adherence.

The investigators propose to develop and validate MyRareDiet® (MRD) to address an unmet need in the IEM population to assist with dietary tracking while facilitating the collection of dietary data from individuals with IEM for research purposes. MRD includes a Patient Portal, a Clinical Dietician Portal, and a Researcher Portal. The Patient Portal is to help IEM patients track and monitor their own diet so they can achieve their strict diet targets. The main features include the integration of a major food database for regular foods with a third database for medical foods, the recording of food intake, and daily dietary reports for food monitoring. The Clinical Dietician Portal helps clinical dieticians manage diet modifications for individuals with IEM. It allows a dietitian to individualize MRD for a specific patient based on findings from their nutrition assessment, and set their nutrient goals and restrictions. The Researcher Portal will facilitate the conduct of diet-based studies and the analysis of study results. It offers typical clinical trial management features such as site and staff management, protocol specification, recruitment status, and study data exports.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with urea cycle disorder, propionic acidemia, maple syrup urine disease or methylmalonic acidemia
* consuming a diet where ≥50% of energy is supplied by foods consumed orally
* self-known (or prescribed) dietary energy goal and protein restriction
* internet connected device to access MyRareDiet

Exclusion Criteria:

* pregnant

Ages: 1 Year to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11-15 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Energy | 24 hour
  Total reported energy intake
Protein | 24 hour
  Total percent of calories from protein

SECONDARY OUTCOMES:
Carbohydrate | 24 hour
  total percent of calories from carbohydrate
Fat | 24 hour
  Total percent of calories from Fat

CONTACTS AND LOCATIONS:
Overall Officials: Dershung Yang, PhD, Principal Investigator — BrightOutcomes, Inc.

IPD SHARING:
Plan to Share IPD: No
The confidentiality of subjects' data will be maintained by use of de-identification procedures. Informed consent forms that include the subject's name will be stored separately in locked file cabinets. Electronic records will be handled according to HIPAA rules where individually identifiable data, such as names, any identification numbers and certain demographic information, are stored separately and password-protected so that they can be accessed only by the project Investigators. A unique subject identifier (ID) will be generated for each participant and used by the subject to access the developed prototype system and for researchers to retrieve information related to a specific subject. At the end of this study, all patient identifiable data in all formats will be completely destroyed.